CLINICAL TRIAL: NCT00089362
Title: Phase 1 Study of 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG, NSC #707545) in Patients With Solid Tumors.
Brief Title: Alvespimycin Hydrochloride in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01455; 04-053; MSKCC-04053; NCI-6542; CDR0000378288; U01CA069856 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Male Breast Cancer; Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Basal Cell Carcinoma of the Lip; Recurrent Breast Cancer; Recurrent Colon Cancer; Recurrent Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Recurrent Gastric Cancer; Recurrent Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Recurrent Lymphoepithelioma of the Nasopharynx; Recurrent Lymphoepithelioma of the Oropharynx; Recurrent Melanoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Ovarian Epithelial Cancer; Recurrent Prostate Cancer; Recurrent Renal Cell Cancer; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Basal Cell Carcinoma of the Lip; Stage III Colon Cancer; Stage III Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage III Gastric Cancer; Stage III Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage III Lymphoepithelioma of the Nasopharynx; Stage III Lymphoepithelioma of the Oropharynx; Stage III Melanoma; Stage III Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Ovarian Epithelial Cancer; Stage III Renal Cell Cancer; Stage III Salivary Gland Cancer; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Nasopharynx; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Adenoid Cystic Carcinoma of the Oral Cavity; Stage IV Basal Cell Carcinoma of the Lip; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Esthesioneuroblastoma of the Paranasal Sinus and Nasal Cavity; Stage IV Gastric Cancer; Stage IV Inverted Papilloma of the Paranasal Sinus and Nasal Cavity; Stage IV Lymphoepithelioma of the Nasopharynx; Stage IV Lymphoepithelioma of the Oropharynx; Stage IV Melanoma; Stage IV Midline Lethal Granuloma of the Paranasal Sinus and Nasal Cavity; Stage IV Mucoepidermoid Carcinoma of the Oral Cavity; Stage IV Ovarian Epithelial Cancer; Stage IV Prostate Cancer; Stage IV Renal Cell Cancer; Stage IV Salivary Gland Cancer; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity; Unspecified Adult Solid Tumor, Protocol Specific; Untreated Metastatic Squamous Neck Cancer With Occult Primary
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms; Colonic Neoplasms; Esthesioneuroblastoma, Olfactory; Stomach Neoplasms; Melanoma; Carcinoma, Ovarian Epithelial; Prostatic Neoplasms; Carcinoma, Renal Cell; Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — 17-(dimethylaminoethylamino)-17-demethoxygeldanamycin

ARMS (1):
- Treatment (alvespimycin hydrochloride) (Experimental): Patients receive alvespimycin hydrochloride IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 1-2 patients receive accelerated escalating doses of alvespimycin hydrochloride until at least 1 of 2 patients experience DLT. Cohorts are then expanded to 3-6 patients who receive escalating doses (in a standard manner) of alvespimycin hydrochloride until MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT. Once the MTD is determined, 10 additional patients are treated at that dose.
  Interventions: Drug: alvespimycin hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: alvespimycin hydrochloride — Given IV
  Other Names: 17-DMAG HCL; KOS-1022
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of alvespimycin hydrochloride in treating patients with metastatic or unresectable solid tumors. Drugs used in chemotherapy, such as alvespimycin hydrochloride, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxic effects and maximum tolerated dose of 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) in patients with metastatic or unresectable solid tumors.

SECONDARY OBJECTIVES:

II. Determine the effects of this drug on the expression of Hsp90 client proteins in normal and tumor tissue samples from these patients.

OUTLINE: This is a dose-escalation study.

Patients receive alvespimycin hydrochloride IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-2 patients receive accelerated escalating doses of alvespimycin hydrochloride until at least 1 of 2 patients experience dose-limiting toxicity (DLT). Cohorts are then expanded to 3-6 patients who receive escalating doses (in a standard manner) of alvespimycin hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience DLT. Once the MTD is determined, 10 additional patients are treated at that dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor, including, but not limited to, the following:

  * Prostate
  * Breast
  * Ovary
  * Colon
  * Kidney
  * Head and neck
  * Stomach
  * Melanoma
* Metastatic or unresectable disease
* No standard curative or palliative therapy exists or is no longer effective
* Progressive disease as indicated by the following:

  * Non-prostate cancer

    * New lesions or increase in pre-existing lesions on bone scintigraphy, CT scan, MRI, or by physical examination
    * No increase in biochemical markers (e.g., carcinoembryonic antigen or CA-15-3) or symptoms as sole evidence of disease progression
  * Prostate cancer

    * Must have castrate metastatic disease (i.e., disease progression after castration or treatment with a gonadotropin-releasing hormone [GnRH] analog)

      * Patients who have not undergone surgical orchiectomy must continue with medical therapy (i.e., GnRH analogs) to maintain castrate levels of serum testosterone < 50 ng/dL
      * Patients who received an antiandrogen as part of first-line hormonal therapy must show disease progression after discontinuing treatment
    * Progressive metastatic disease on imaging studies (e.g., bone scan, CT scan, or MRI) OR metastatic disease and a rising prostate-specific antigen (PSA) allowed

      * Biochemical progression is defined as a minimum of 3 rising PSA values from baseline obtained at least 1 week apart OR 2 rising PSA values obtained more than 1 month apart, with >= 25% increase in value
* No active brain metastases
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - Karnofsky 70-100%
* Performance status - ECOG 0-1
* More than 6 months
* WBC >= 3, 000/mm^3
* Absolute neutrophil count >= 1, 500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* AST and ALT < 1.5 times ULN
* PT normal
* Creatinine =< 1.4 mg/dL
* Creatinine clearance > 55 mL/min
* QTc < 450 msec for male patients (470 msec for female patients)
* LVEF > 40% by MUGA
* No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation >= 3 beats in a row)
* No myocardial infarction within the past year
* No active ischemic heart disease within the past year
* No New York Heart Association class III or IV congestive heart failure
* No congenital long QT syndrome
* No left bundle branch block
* No poorly controlled angina
* No history of uncontrolled dysrhythmias or requiring antiarrhythmic drugs

  * Calcium blockers and beta blockers allowed
* No other significant cardiac disease
* Oxygen saturation > 88%
* Dyspnea < grade 2 at rest on room air
* No clinically significant pulmonary comorbidity (e.g., severe chronic obstructive pulmonary disease)
* No requirement for supplemental oxygen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active or ongoing infection
* No symptomatic peripheral neuropathy >= grade 2
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin and nitrosoureas)
* At least 1 week since prior ketoconazole
* More than 4 weeks since prior radiotherapy
* Recovered from all prior therapy
* More than 4 weeks since prior investigational anticancer therapeutic drugs
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent administration of any of the following herbal remedies:

  * Hydrastis canadensis (goldenseal)
  * Hypericum perforatum (St. John's wort)
  * Uncaria tomentosa (cat's claw)
  * Echinacea angustifolia roots
  * Trifolium pratense (wild cherry)
  * Matricaria chamomilla (chamomile)
  * Glycyrrhiza glabra (licorice)
  * Dillapiol
  * Hypericin
  * Naringenin
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
MTD, defined as the dose level where the observed DLT incidence in no more than one out of six patients treated at a particular dose level | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: David Solit, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States